CLINICAL TRIAL: NCT06065215
Title: Early-life MRI Biomarkers of Longer-term Respiratory Morbidity in Infants Born Extremely Preterm (EMBLEM)
Acronym: EMBLEM
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: The Hospital for Sick Children (Other); MOUNT SINAI HOSPITAL (Other); Hannover Medical School (Other); St. Justine's Hospital (Other); Montreal Children's Hospital of the MUHC (Other)
Responsible Party: Principal Investigator, Sherri Katz, Division Head, Senior Scientist, Pediatric Respirologist, Children's Hospital of Eastern Ontario
Other Study IDs: 486713
Record Dates: First submitted 2023-09-27; First posted 2023-10-03 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Lung Function; BPD - Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Magnetic Resonance Imaging; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging (MRI) — Magnetic Resonance Imaging (MRI) is a non-invasive medical imaging technique that uses powerful magnets and radio waves to generate detailed images of the body's internal structures. The MRI intervention includes using a specialized MRI machine and lung imaging protocol.
Diagnostic Test: Echocardiogram — An echocardiogram, often called an "echo," is a non-invasive medical test that uses high-frequency sound waves (ultrasound) to create real-time images of the heart's structure and function. It provides valuable information about the heart's size, shape, and function.
Diagnostic Test: Lung ultrasound — Lung ultrasound is a non-invasive imaging technique that employs high-frequency sound waves (ultrasound) to visualize the structures and conditions of the lungs. It is particularly valuable for diagnosing and monitoring lung-related conditions, such as pneumonia, pleural effusions, and pulmonary edema. The lung ultrasound intervention involves using an ultrasound machine equipped with a specialized probe gently placed on the chest to capture detailed images of the lungs and adjacent structures.

SUMMARY:
Bronchopulmonary dysplasia (BPD) is a common, major complication of premature birth, associated with developmental and health consequences that continue into adulthood. Prediction of who will have these problems is challenging using traditional definitions of disease. It is believed that underdevelopment and injury occur in both lung tissue and the blood vessels in the lungs, with a sophisticated interplay between them that contributes to lung disease seen in prematurity. New magnetic resonance imaging (MRI) techniques can delineate tissue structure with unprecedented granularity, assessing lung tissue, blood vessels, and their interplay. The ability to identify, at an early stage, those infants destined for chronic lung disease with greater certainty will be useful in counseling families and critical for the effective introduction of promising new BPD therapies. 319 infants born less than 29 weeks gestation will be recruited from 4 centres, including 5 babies who received stem cell therapy in a clinical trial. Babies will be evaluated at 36 weeks post-conception with lung MRI, oscillometry (lung function), echocardiogram (heart ultrasound), and oscillometry. Lung health will be assessed every 3 months by phone questionnaire and chart review. At 18-21 months post-conception, babies will undergo neurodevelopmental assessment and lung function testing. The investigators will look at how well baseline MRI markers predict subsequent lung health and development, independently and combined with echocardiogram, lung ultrasound, and traditional markers of BPD. The investigators anticipate that these new MRI markers will measure lung health safely and longitudinally in babies born extremely preterm. By identifying predictors of longer-term lung disease, clinicians will be able to allocate resources to babies at the highest risk of severe disease. Further, The investigators envision that MRI will help identify babies who would benefit most from interventions like stem cell therapy and be useful for evaluation of future treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born at <29 weeks gestation;
2. currently <36 weeks PMA.

Exclusion Criteria:

1. Known interstitial lung disease, congenital lung anomaly, ciliary dysfunction, immunodeficiency, cystic fibrosis, neuromuscular disease, or structural heart disease (other than atrial septal defect/hemodynamically insignificant ventricular septal defect/patent ductus arteriosus);
2. genetic syndrome or congenital anomaly;
3. contraindications for MRI or transport;
4. invasive or non-invasive ventilation that cannot be safely removed for MRI;
5. current respiratory infection;
6. family cannot speak English/French;
7. transferred to another hospital prior to baseline study visit
8. not receiving follow-up at one of the study centres.

Ages: 35 Weeks to 21 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Babies will be recruited from four Canadian tertiary care pediatric centers: Children's Hospital of Eastern Ontario (CHEO), Ottawa, ON; Mount Sinai Hospital, Toronto, ON; Centre Hospitalier Universitaire Sainte-Justine, Montreal QC; and Montreal Children's Hospital, Montreal QC. MRI will occur at each site except Mount Sinai, whose babies will undergo MRI at The Hospital for Sick Children, Toronto, ON.
Sampling Method: Non-Probability Sample
Enrollment: 319 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Severe Post-prematurity Respiratory Disease (PRD) | The evaluation will be conducted at regular intervals of every 3 months, commencing at 36 weeks PMA and continuing until the child reaches 18 months corrected age
  PRD will be defined based on the consensus definition of the Prematurity and Respiratory Outcomes Program. This composite outcome characterizes clinically relevant persistent respiratory morbidity in early life. It will be evaluated every 3 months from 36 weeks PMA to 18 months corrected age through parent questionnaire and chart review. Severe PRD is defined as a positive response to any of the following: ≥2 respiratory-related hospitalizations, home oxygen at 3 months corrected age or any home respiratory support, systemic corticosteroid or pulmonary vasodilators after discharge home, chronic respiratory symptoms (cough without cold or wheeze at least once per week) despite concurrent inhaled corticosteroids in ≥ 2 questionnaires, or death secondary to a cardiopulmonary cause. PRD has been used as a clinical outcome in cohort studies and an American Thoracic Society guideline on optimal neonatal care pathways and predictive perinatal characteristics.

SECONDARY OUTCOMES:
Neurodevelopmental Impairment (NDI) | Neurodevelopmental impairment will be determined at the 18-21 months corrected age visit
  Per the Canadian Neonatal Follow-Up Network protocol, NDI will be determined at the 18-21 months corrected age visit. Children will be administered the Bayley Scales of Infant and Toddler Development, 4th edition (Bayley-4), assessing infant developmental functioning across five domains. Cognition, language, and motor subtests are directly assessed by a blinded, trained assessor regarding neonatal history. The social-emotional and adaptive behavior components are assessed via parental questionnaires. The Bayley-4 yields standard mean scores of 100±15. A pediatrician performs a neurological examination to identify signs of cerebral palsy and determine functional level using the Gross Motor Functional Classification System (GMFCS). Visual and hearing function data are retrieved from the chart. NDI will be defined as the presence of any of the following: Bayley-4 score <85, cerebral palsy with GMFCS ≥ 2, the requirement for hearing aids/cochlear implants, and bilateral blindness.

CONTACTS AND LOCATIONS:
Overall Officials: Sherri Katz, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (4):
- Canada (4):
  - The Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - CHU-Sainte Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No